CLINICAL TRIAL: NCT01207310
Title: Pager-Assisted Smoking Cessation Treatment
Acronym: Pager
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Timothy Carmody, Health Sciences Clinical professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11RT0009
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Smoking Cessation
Keywords: smoking; smoking of 10 cigarettes per day
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Behavior Therapy; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pager Arm (Experimental): Participants in the Pager Arm will be provided with alphanumeric pagers and will receive therapeutic messages on these pagers for 3 months in addition to individual smoking cessation counseling and nicotine patches.
  Interventions: Behavioral: smoking cessation counseling; Drug: Nicotine patch; Device: alphanumeric pager
- Control Arm (Active Comparator): Participants in the Control Arm will receive individual smoking cessation counseling and nicotine patches.
  Interventions: Behavioral: smoking cessation counseling; Drug: Nicotine patch

INTERVENTIONS:
Behavioral: smoking cessation counseling — two 60-minute face-to-face treatment sessions and three 20-minute follow-up contacts at weeks 2, 3, and 9
  Other Names: Behavioral counseling
Drug: Nicotine patch — 8 weeks' worth of nicotine patches
  Other Names: Nicoderm
Device: alphanumeric pager — therapeutic messages to be delivered for three months
  Other Names: Pager-assisted text messaging
  Arms: Pager Arm

SUMMARY:
The proposed study tests the efficacy of using pager-assisted messages combined with nicotine patches in facilitating smoking cessation and relapse prevention in a 2-arm randomized clinical trial. The hypothesis is that the proportion of biochemically-verified quitters at 3 and 12 months in the study arm randomized to receive therapeutic messages on alphanumeric pagers for 3 months along with individual smoking cessation counseling and nicotine patches will be greater that the proportion of biochemically-verified quitters who receive only individual smoking cessation counseling and nicotine patches.

DETAILED DESCRIPTION:
A total of 224 current smokers were enrolled in a randomized controlled smoking cessation trial. Participants were community-living adult smokers of ≥10 cigarettes per day during the pre-enrollment week who were interested in quitting and recruited from the local area by means of print, media, and online advertisements. To be eligible, they needed to be smoking 10 or more cigarettes per day, aged 18 or older, motivated to quit smoking, prepared to set a quit date, willing to use nicotine patches, and able to come to therapy sessions and be followed by telephone. Participants in the pager treatment were provided with alpha-numeric pagers free of charge for three months. Using specially-designed communication software, text messages were sent to participants aimed at facilitating motivation to quit, cessation strategies, and coping skills to maintain abstinence. Participants in both treatment groups were seen for two 60-minute sessions of standard smoking cessation counseling, and received three follow-up phone calls and two months of nicotine patches.

ELIGIBILITY:
Inclusion Criteria:

* smoking 10 or more cigarettes per day
* aged 18 or older
* motivated to quit smoking and prepared to set a quit date
* willing to use nicotine patches
* ability to come to therapy sessions and be followed by telephone

Exclusion Criteria:

* individuals who are psychotic
* severely depressed
* organically brain impaired
* actively abusing alcohol or other substances, and/or who have been drug dependent during the past six months
* terminally ill
* unable to be contacted by phone,currently using nicotine replacement or smoking cessation medications
* those with contraindications to nicotine patches, female smokers who are pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2003-05; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
biologically-validated point prevalence smoking cessation | 12 months after enrollment
  Abstinence from cigarettes "even a puff", other tobacco products and nicotine replacement for seven days at the 12 month follow-up date as validated by salivary cotinine less than 15 ng/ml

SECONDARY OUTCOMES:
continuous abstinence from cigarettes "even a puff", tobacco products and nicotine replacement | 12 months after enrollment
  maintained cessation from smoking, biologically-validated by repeated measures of salivary cotinine less than 15 ng/ml at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy P Carmody, Ph.D, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Veterans Affairs Medical Center, San Francisco, California, United States